CLINICAL TRIAL: NCT01098149
Title: Tolerance to Hemodialysis in Insulin-Requiring Diabetic Patients: a Prospective Randomized,Cross-over Multicenter Study Between Bicarbonate Dialysis (BD) and Blood Volume Controlled Acetate-Free Biofiltration (BVC-AFB)
Brief Title: Tolerance to Hemodialysis in Insulin-Requiring Diabetic Patients: BD vs AFB With Blood Volume Biofeedback
Acronym: THIRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Dott.Ezio Movilli, Dept of Nephrology -Brescia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: THIRD-01
Record Dates: First submitted 2010-03-29; First posted 2010-04-02 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Hypotension; Hemodialysis
Keywords: Haemodialysis treatment tolerance; acetate free biofiltration; frequency of hypotensive events during dialysis; nurse intervention during dialysis
MeSH Terms: conditions — Hypotension | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AFB stand alone (Active Comparator): Patients are switched in AFB treatment, without blood volume control.
  Interventions: Other: BD and BVC, AFB
- BD and BVC (Active Comparator): Patients are switched into bicarbonate dialysis with Blood Volume Control
  Interventions: Other: BD and BVC, AFB

INTERVENTIONS:
Other: BD and BVC, AFB — Some patients are randomized into the AFB, the others into the BD and BVC
  Other Names: Biofeedback,Blood Volume Control,Acetate Free Biofiltration

SUMMARY:
Diabetic nephropathy is becoming the most common primary renal disease in end stage renal disease patients. The prevalence of diabetic patients in dialysis reaches even the 30% of the dialysis population (USRDS) with an incidence rate, in some countries, up to 40%. The 5 years surviving time of diabetic patients in dialysis is about the 20% and, compared to the hypertension and glomerulonephritis complications, still remains the worst. Diabetes is often associated to several comorbid factors such as hypertension, autonomic neuropathy, vasculopathy, metabolic disorders (ketoacidosis, poor glycaemic control), and electrolyte disorders. So, the diabetic patient is fragile, with a rather poor tolerance to dialysis, lack of achievement of dry body weight and inadequate dialysis. In order to gain a more detailed insight into a possible better tolerance to dialysis, arising from the elimination of acetate in dialysate bath (Acetate Free Biofiltration) and from the use of an automatic system to control the blood volume (Blood Volume Control),the investigators would like to investigate the cardiovascular stability and the frequency of intradialytic symptoms in a prospective, randomized, cross-over study.

DETAILED DESCRIPTION:
Acetate-Free-Biofiltration (AFB) was proved to be a technique suitable to treat critical patients, such as elders and diabetics, because of frequency reduction of hypotensive episodes and symptoms during the treatment and a better control to metabolic aspects (such as metabolic acidosis).

The Blood Volume Control (BVC) is a tool, that allows to improve the cardiovascular tolerance to the treatment, especially in hypotension-prone patients, appearing promising in the correction of the arterial hypertension induced by the hydro-saline overload.

The use of BVC in AFB has been tested to verify the behaviour of the kinetics of electrolyte (in particular of bicarbonate) and it has got good results, in terms of a further improvement in treatment tolerance, for critical patients However, this therapy (AFB+BVC) was not yet evaluated as the dialysis tolerance improvement in diabetics concern, nor the relative contribution given by each factor in achieving this result.

The study, 9 months long, is aimed to verify the treatment tolerance of insulin requiring diabetic patients, by using standard bicarbonate dialysis (BD), or Acetate Free Biofiltration (AFB) and/or a Blood Volume Control(BVC). The study is divided in three phases: the first one, three months long, is the baseline in standard bicarbonate dialysis, then all the patients are shifted to AFB with BVC, for other three months, while the last three months long phase, after a randomization, has the aim to identify the relative contribution of each factor (absence of acetate in the bath or BVC) in the treatment tolerance improvement(if any). The treatment tolerance will be evaluated considering the frequency of intradialytic hypotensive events.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease patients
* Patients affected by diabetic nephropathy with insulin therapy, for, at least, 6 months
* Patients with renal replacement therapy with haemodialysis three time a week, for, at least, 6 months.
* Age between 18 and 85 years

Exclusion Criteria:

* Patients affected by neoplasm and/or mental illness
* Patients with residual diuresis > 500 ml/die;
* Patients in single needle bicarbonate dialysis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Investigate a possible better tolerance to dialysis, eliminating acetate in the dialysate bath, with AFB treatment, and using, at the same time, the automatic blood volume control (BVC). | 3 months
  The treatment tolerance is measured by the number of intradialytic hypotensive events, defined as:
  * systolic blood pressure less then 90 mmHg;
  * systolic blood pressure more then 25 mmHg to the predialysis value, with hypotensive events requiring therapies;
  * systolic blood pressure less then 90 mmHg with hypotensive events requiring therapies for those patients, which predialysis systolic blood pressure value was 100 mmHg.

SECONDARY OUTCOMES:
The secondary outcome measure is to evaluate the relative efficiency of each factor (AFB in the bath and blood volume control) to reach this result. | 3 months
  The evaluation will be done on:
  * frequency of hypotensive events, during dialysis (defined as above);
  * number of nurse interventions (defined as ultrafiltration rate stop, or saline infusion);
  * antihypertensive drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Cancarini, MD, Study Chair — Università of Brescia
Locations (5):
- Italy (5):
  - Hospital "Santa Maria della Scaletta", Imola, Bologna
  - Hospital "Nuovo Ronco", Gussago, Brescia
  - Hospital "Policlinico S.Orsola-Malpighi", Bologna
  - Hospital "Spedali Civili", Brescia
  - Hospital "Degli Infermi", Rimini

REFERENCES:
- [Background] Movilli E, Camerini C, Zein H, D'Avolio G, Sandrini M, Strada A, Maiorca R. A prospective comparison of bicarbonate dialysis, hemodiafiltration, and acetate-free biofiltration in the elderly. Am J Kidney Dis. 1996 Apr;27(4):541-7. doi: 10.1016/s0272-6386(96)90165-1. PMID 8678065
- [Background] Verzetti G, Navino C, Bolzani R, Galli G, Panzetta G. Acetate-free biofiltration versus bicarbonate haemodialysis in the treatment of patients with diabetic nephropathy: a cross-over multicentric study. Nephrol Dial Transplant. 1998 Apr;13(4):955-61. doi: 10.1093/ndt/13.4.955. PMID 9568857
- [Background] Santoro A, Mancini E, Basile C, Amoroso L, Di Giulio S, Usberti M, Colasanti G, Verzetti G, Rocco A, Imbasciati E, Panzetta G, Bolzani R, Grandi F, Polacchini M. Blood volume controlled hemodialysis in hypotension-prone patients: a randomized, multicenter controlled trial. Kidney Int. 2002 Sep;62(3):1034-45. doi: 10.1046/j.1523-1755.2002.00511.x. PMID 12164888
- [Background] Ronco C, Brendolan A, Milan M, Rodeghiero MP, Zanella M, La Greca G. Impact of biofeedback-induced cardiovascular stability on hemodialysis tolerance and efficiency. Kidney Int. 2000 Aug;58(2):800-8. doi: 10.1046/j.1523-1755.2000.00229.x. PMID 10916105